CLINICAL TRIAL: NCT04726709
Title: Alexander Technique Classes - Multisite
Brief Title: Poised for Parkinson's - an Intervention to Increase Embodied Agency in People With Parkinson's Disease and Their Carers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Idaho (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Rajal Cohen, Associate Professor, University of Idaho
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-164; U54GM104944 (NIH)
Record Dates: First submitted 2021-01-12; First posted 2021-01-27 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Parkinson's Disease
Keywords: Alexander Technique; Posture; Mindfulness; Embodiment; Caregivers; Movement Interventions; Complementary Integrative Medicine; Non-pharmacological interventions; Quality of Life
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Poised for Parkinson's (Experimental): Alexander-technique-based online course to increase embodied agency in people with Parkinson's disease and their care partners.
  Interventions: Behavioral: Poised for Parkinson's

INTERVENTIONS:
Behavioral: Poised for Parkinson's — Lecture, demonstration, activities, and supplemental materials designed to improve self-awareness, situational awareness, and ability to make good choices for physical and emotional self-care, moment-to-moment.

SUMMARY:
The purpose of the study is to develop, deliver, and test an online Alexander-based training program for people with Parkinson's disease and their care partners.

DETAILED DESCRIPTION:
Six dyads, each consisting of a person with Parkinson's disease and their care partner, will participate in a real-time online course called "Poised for Parkinson's." The course will meet twice per week via Zoom for eighteen 105-minute sessions. Outcome measures, including surveys, interviews, balance, and motor performance, will be assessed the week before classes begin and the week after classes end.

ELIGIBILITY:
Inclusion Criteria:

* dyad including care partner and person with Parkinson's disease
* Hoehn & Yahr Stage 2 (estimated)
* vision and hearing (corrected to) normal
* able to use computer, Internet, and Zoom
* ambulatory without assistive devices
* reside in Idaho

Exclusion Criteria:

* dementia (screen with MOCA)
* severe musculoskeletal pain (screen in interview)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2022-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Poise Project, Candler, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual data will be made available on request.
Supporting Information: Study Protocol, ICF
Time Frame: For five years, starting upon publication
Access Criteria: upon request: email PI. rcohen@uidaho.edu

REFERENCES:
- See also: The Poise Project is delivering the intervention — https://www.thepoiseproject.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited through emails to support group leaders, church leaders, offices of aging, and in-person connections from attendance at pre-COVID Parkinson's events.
Pre-assignment Details: We did not exclude any enrolled participants. One dyad (two participants) dropped out before initial data collection due to discomfort with technology. Numbers in table refer to participants, not dyads.
Groups:
- Poised for Parkinson's - Patients: Alexander-technique-based online course to increase embodied agency in people with Parkinson's disease and their care partners.
  Poised for Parkinson's: Lecture, demonstration, activities, and supplemental materials designed to improve self-awareness, situational awareness, and ability to make good choices for physical and emotional self-care, moment-to-moment.
- Poised for Parkinson's - Care Partners: Alexander-technique-based online course to increase embodied agency in people with Parkinson's disease and their care partners.
Period: Overall Study
Arm/Group | Poised for Parkinson's - Patients | Poised for Parkinson's - Care Partners
Started | 16 | 14
Completed | 14 (These numbers refer to individual participants, not dyads.) | 12
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Poised for Parkinson's - Patients: Alexander-technique-based online course to increase embodied agency in people with Parkinson's disease and their care partners.
  Poised for Parkinson's: Lecture, demonstration, activities, and supplemental materials designed to improve self-awareness, situational awareness, and ability to make good choices for physical and emotional self-care, moment-to-moment.
  Outcome measures specific to patients include surveys of symptom self-management and objective assessments of physical performance and balance.
- Poised for Parkinson's - Care Partners: Alexander-technique-based online course to increase embodied agency in people with Parkinson's disease and their care partners.
  Poised for Parkinson's: Lecture, demonstration, activities, and supplemental materials designed to improve self-awareness, situational awareness, and ability to make good choices for physical and emotional self-care, moment-to-moment.
  Outcome measures specific to care partners include surveys of care recipient symptom self-management.
- Total: Total of all reporting groups
Arm/Group | Poised for Parkinson's - Patients | Poised for Parkinson's - Care Partners | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 12 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (8.4) | 67.6 (6.7) | 68.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 11 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 14 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Motor Function - Objective
Description: Physical Performance Test (7 items). Score can vary from 0-28. Higher score is better.
Time Frame: Assessed the week before the intervention (week 1) and the week after the intervention (week 11). Difference is reported. Positive number indicates improvement.
Population: Participants included people with PD and their care partners. Only people with PD were assessed with objective measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Poised for Parkinson's - Patients
Number analyzed (Participants) | 14
score on a scale | 0.93 (2.16)

2. Primary Outcome: Balance - Objective
Description: Due to COVID, we only assessed the subset of brief Bestest that can be scored online: standing on each foot, gait stability, and forward reach. Possible scores: 0-12. Higher score is better. Positive number indicates improvement.
Time Frame: as for outcome 1
Population: Only participants with PD are included in this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Poised for Parkinson's
Number analyzed (Participants) | 14
score on a scale | 0.43 (1.65)

3. Primary Outcome: Balance: Self-report
Description: Activities Balance Confidence scale. Possible score from 0-100. Higher score is better.
Time Frame: as for outcome 1
Population: Only people with PD were assessed with this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Poised for Parkinson's
Number analyzed (Participants) | 14
score on a scale | 2.9 (11.9)

4. Primary Outcome: Posture - Objective
Description: Assessed by photo in sagittal plane. Positive numbers indicate a more upright posture.
Time Frame: as for outcome 1
Population: Only participants with PD were assessed.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Poised for Parkinson's
Number analyzed (Participants) | 14
degrees | 2.0 (6.7)

5. Secondary Outcome: Feasibility - Attendance
Description: Course attendance (out of 16)
Time Frame: Attendance will be tracked at every class session, weeks 2-10.
Population: people with Parkinson's disease
Measure: Mean (Standard Deviation); unit: number of classes attended
Arm/Group | Poised for Parkinson's
Number analyzed (Participants) | 14
number of classes attended | 14.2 (3.8)

6. Secondary Outcome: Feasibility - Retention
Description: Study retention: number of participants who completed the study
Time Frame: assessed after the intervention (week 11)
Population: both participants with PD and care partners
Measure: Count of Participants; unit: Participants
Groups:
- People Living With Parkinson's Disease: Alexander-technique-based online course to increase embodied agency in people with Parkinson's disease and their care partners.
- Care Partners: People living with Parkinson's disease and their care partners normally attend class together, but it is possible that one might complete the class and the other might not.
Arm/Group | People Living With Parkinson's Disease | Care Partners
Number analyzed (Participants) | 16 | 14
Participants | 14 | 12

7. Secondary Outcome: Symptom Management
Description: Survey administered by phone, with 29 Likert scale questions on a scale of 0-5 asking how well the person with Parkinson's disease is able to manage typical Parkinson's symptoms, including bradykinesia, tremor, stooped posture, freezing of gait, anxiety, fatigue, and so on. Higher scores indicate better symptom management. The scores were summed, with a possible range of 0-145.
Time Frame: as for outcome 1
Population: self-report from people with PD
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Poised for Parkinson's
Number analyzed (Participants) | 14
units on a scale | 10.14 (12.20)

8. Secondary Outcome: Care-partner Self-management Skill
Description: Anonymous course evaluation survey filled out and mailed in. Question reported: I feel I am better prepared for the present and future daily challenges of being my partner's care partner. Rate from 1-10 with 10 being high.
Time Frame: Assessed after the intervention (week 11)
Population: Only care partners were asked this question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Poised for Parkinson's - Care Partners
Number analyzed (Participants) | 12
units on a scale | 8.7 (1.9)

ADVERSE EVENTS:
Time Frame: 4 months
Description: There were no adverse events.
Arm/Group | Poised for Parkinson's - Patients | Poised for Parkinson's - Care Partners
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

LIMITATIONS AND CAVEATS:
Study conducted during COVID. All assessments conducted via Zoom.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT04726709/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT04726709/ICF_001.pdf